CLINICAL TRIAL: NCT01909687
Title: Leistungsbewertung Von Blutzuckermesssystemen im Methodenvergleich
Brief Title: Assessment of Blood Glucose Monitoring Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: IDT-1313-SF
Record Dates: First submitted 2013-07-02; First posted 2013-07-26 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes
Keywords: blood glucose monitoring systems; ISO 15197; system accuracy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Blood glucose monitoring systems
  Other Names: Accu-Chek Aviva; Contour XT; FreeStyle Insulinx; Accu-Chek Performa; Contour next USB; BGStar; OneTouch Verio IQ; MyStar Extra; mylife Pura; Glucocard G+

SUMMARY:
System accuracy evaluation of different blood glucose monitoring systems with 3 lots of test strips per systems according to ISO 15197:2013

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Male or female subjects with type 1 or type 2 diabetes or healthy subjects
* For BG adjustment people with type 1 diabetes

Exclusion Criteria:

* Severe acute illness that, in the opinion of the Investigator, might pose additional risk to the patient
* Chronic illness that, in the opinion of the Investigator, might pose additional risk to the patient
* Current condition that, in the opinion of the Investigator, doesn't enable subject to participate in the study
* For BG adjustment people with type 1 diabetes without CHD, condition after myocardial infarction, PAOD, cerebral events or hypoglycaemia unawareness
* Legal incompetence or limited legal competence
* Age < 18 years
* Dependency from the sponsor or the clinical investigator
* Mental incapacity or language barriers precluding adequate compliance with the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Analysis of system accuracy | for each subject, the experimental phase has an expected duration of up to 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft an der Universität Ulm, Ulm, Germany

REFERENCES:
- [Result] Freckmann G, Link M, Schmid C, Pleus S, Baumstark A, Haug C. System Accuracy Evaluation of Different Blood Glucose Monitoring Systems Following ISO 15197:2013 by Using Two Different Comparison Methods. Diabetes Technol Ther. 2015 Sep;17(9):635-48. doi: 10.1089/dia.2015.0085. Epub 2015 Jun 25. PMID 26110670